CLINICAL TRIAL: NCT06039969
Title: Study on the Changes of Intestinal Flora and Cardiac Fibrosis in Patients With Dilated Cardiomyopathy Diagnosed for the First Time by Sports Rehabilitation
Brief Title: Evaluate Aerobic Exercise on Myocardial Fibrosis and Intestinal Flora in Dilated Cardiomyopathy Diagnosed First Time.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jin Geng, associate doctor, Nanjing Medical University
Other Study IDs: 20230911
Record Dates: First submitted 2023-09-11; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Cardiac Rehabilitation; Myocardial Fibrosis
Keywords: Aerobic exercise rehabilitation; Myocardial Fibrosis; human gut microbiome; cardiac magnetic resonance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cardiac MRI data and patient's feces will be collected.Changes in intestinal flora spectrum will be detected.

GROUPS / COHORTS (1):
- Cardiac MRI will be performed in patients with heart failure caused by cardiomyopathy.: Cardiac MRI will be performed in patients with heart failure caused by cardiomyopathy. At the same time Collect patient feces.this is a obvertional study ,ther is no intervetion

INTERVENTIONS:
Other:  — This is an obvertional study and there is no intervention

SUMMARY:
To invegstive the Changes of Intestinal Flora and the improvements of Cardiac Fibrosis in Patients With Dilated Cardiomyopathy Diagnosed for the First Time by heart Rehabilitation

DETAILED DESCRIPTION:
Previous studies have confirmed that Aerobic exercise rehabilitation can reduce the rate of readmission of patients with heart failure and improve their cardiopulmonary endurance and exercise ability. However, whether aerobic exercise rehabilitation can inhibit myocardial fibrosis or delay the progress of fibrosis in patients with heart failure has not been reported. At the same time, some studies have shown that the change of intestinal microbial flora may promote the progress of heart failure, and regular aerobic exercise will also lead to the change of intestinal microbial flora, but whether aerobic exercise rehabilitation can improve intestinal microbial flora in patients with dilated cardiomyopathy has not been reported. In our study, patients who were hospitalized for heart failure for the first time and were finally diagnosed with dilated cardiomyopathy were recruited. Recruited patients will enter the routine cardiac rehabilitation process and make an individualized aerobic exercise plan according to the cardiopulmonary exercise test. Cardiac MRI and intestinal microflora changes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 1、Patients hospitalized for the first time because of heart failure 2、The patient who was definitely diagnosed as dilated cardiomyopathy for the first time

Exclusion Criteria:

* 1、Other types of cardiomyopathy 2、Has been diagnosed as dilated cardiomyopathy. 3、malignant tumor 4、acute infection 5、Cannot perform cardiopulmonary exercise test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were hospitalized for heart failure for the first time and were finally diagnosed with dilated cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
myocardial fibrosis | first admission six months one year
  Assessment of myocardial fibrosis based on cardiac MRI examination

SECONDARY OUTCOMES:
Bacterial spectrum of intestine | first admission six months one year
  Assessment of Bacterial spectrum of intestine based on Patient feces sequencing

OTHER OUTCOMES:
cardiac fitiness | first admission six months one year
  Assessment of caridac fitness based on ardiopulmonary exercise test

CONTACTS AND LOCATIONS:
Overall Officials: XiWen Zhang, MD, Study Director — Huai'an First People's Hospital
Locations (1):
- Huai'An First People'S Hospital, Huai'an, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No